CLINICAL TRIAL: NCT05348564
Title: Comparing Direct and Indirect Methods for Cascade Screening in Familial Hypercholesterolemia (FH) and Long QT Syndrome (LQTS)
Brief Title: Comparing Direct vs Indirect Methods for Cascade Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Amber Beitelshees, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R01HL163514 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Long QT Syndrome; Familial Hypercholesterolemia; Ethics; Genetic Testing
MeSH Terms: conditions — Long QT Syndrome; Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct contact (Experimental): Study team contact of family members
  Interventions: Behavioral: Direct contact of family members for cascade screening of relevant variants
- Indirect contact (No Intervention): Proband initiated contact of family members

INTERVENTIONS:
Behavioral: Direct contact of family members for cascade screening of relevant variants — Study team members will directly contact potentially impacted family members to offer genetic testing of relevant variant.
  Arms: Direct contact

SUMMARY:
An important aspect of successful genomic medicine implementation is developing effective approaches for screening at-risk family members after probands are identified, also known as cascade screening. Most cascade screening studies conducted to date have been conducted outside the US, and very few studies have used a rigorous approach involving a comparator group or randomized controlled design. A major question in the field is how to most effectively implement cascade screening, given commonly cited communication barriers, while respecting privacy among probands and family members. This study will conduct a randomized controlled trial to assess direct contact of relatives by study team members vs indirect, or proband-initiated, contact. We will assess efficacy of the cascade screening intervention, patient-centered outcomes regarding mental, physical, and psychosocial outcomes in probands and family members, and implementation evaluation outcomes.

Individuals who are known to carry the KCNQ1 Met224Thr or APOB Arg3527Gln variant will be eligible to participate. After providing consent and being deemed eligible, individuals will be randomized in a 1:1 manner into the direct or indirect contact of family members arm of the study. The randomization will be stratified by variant to ensure equal representation of each variant in the study arms. Individuals in the indirect arm will be instructed to contact their first-degree family members about the opportunity to be screened. They will be provided with a disease-specific pamphlet and a family letter explaining the cascade screening. In the direct arm, probands will be advised that the study staff will be contacting their family members. They will be instructed to also contact their family members prior to the study team contacting them. Approximately two weeks after this meeting with the proband, the study staff will mail letters to eligible first-degree family members of the probands. If we do not hear back from individual family members, we will follow-up with another letter, telephone call, or home visit. The information contained in the letters will be the same information for both the direct and indirect arms of the study. All interested family members will receive pre-test counseling and free, in-home, saliva-based genetic testing, and post-test counseling.

DETAILED DESCRIPTION:
Individuals who are known to carry the KCNQ1 Met224Thr or APOB Arg3527Gln variant will be eligible to participate. After providing consent and being deemed eligible, individuals will be randomized in a 1:1 manner into the direct or indirect contact of family members arm of the study. The randomization will be stratified by variant to ensure equal representation of each variant in the study arms. Individuals in the indirect arm will be instructed to contact their first-degree family members about the opportunity to be screened. They will be provided with a disease-specific pamphlet and a family letter explaining the cascade screening. In the direct arm, probands will be advised that the study staff will be contacting their family members. They will be instructed to also contact their family members prior to the study team contacting them. Approximately two weeks after this meeting with the proband, the study staff will mail letters to eligible first-degree family members of the probands. If we do not hear back from individual family members, we will follow-up with another letter, telephone call, or home visit. The information contained in the letters will be the same information for both the direct and indirect arms of the study. All interested family members will receive pre-test counseling and free, in-home, saliva-based genetic testing, and post-test counseling.

Aim 1:

Aim 1 will assess efficacy of the approaches on uptake of cascade screening. The primary outcome will assess uptake of cascade screening among all first-degree relatives of the probands. We will compare the proportion first-degree relatives who undergo screening out of all eligible relatives in the direct vs indirect arms of the study. Secondary outcomes will asses rate of detection of new cases among all first degree family members. We will have good power to detect a clinically meaningful difference of 15% between he direct and indirect arms of the study.

These cascade screening efficacy endpoints address the question of whether contacting family members for probands improves the uptake of testing among family members.

Aim 2:

Aim 2 will assess patient-centered outcomes in both probands and family members that address how the intervention of direct contact of family members impacts participants' mental, physical, or psychosocial outcomes. For this aim surveys will be given to the probands and family members approximately one week after contact of family members has occurred and at the end of the study. The secondary outcomes associated with this aim include: perceived alignment of ethical principles, anxiety regarding method of contact, perceived pressure to undergo testing (family members only), and knowledge of disease. We will also assess health behaviors such as taking recommended preventative medications (beta-blockers and statins), lifestyle modifications, and seeing health care providers. These outcomes will be assessed by validated and study-created surveys assessed 1-week post implementation and at the end of study.

These patient-centered outcomes assess the extent to which the intervention allows for autonomous decision making and is associated with acceptable psychosocial outcomes.

Aim 3:

Aim 3 will perform qualitative assessments of the intervention to evaluate implementation outcomes in the direct vs indirect arms of the study. We will include interviews among 15 probands randomized to the direct arm, 15 probands randomized to the indirect arm, 15 family members who undergo cascade screening from the direct arm (carriers and non-carriers), 15 family members who undergo cascade screening from the indirect arm (carriers and non-carriers), and 15 family members who decline cascade testing (from direct arm and from indirect arm but informed by a proband, thus allowing us to invite them to participate). We will also interview study staff to understand facilitators and challenges across patient and organizational factors.

Implementation reach, dosage, and fidelity will be based on proportions and means/standard deviations for relevant quantitative variables (e.g., number of genetic counseling visits scheduled and completed). Outreach approach's acceptability, barriers, and facilitators will be based on descriptive analyses using interview data. Data analyses will be based on a codebook, consensus coding and consensus narrative Qualitative interviews will be transcribed verbatim and analyzed using NVivo 11.0. The research team will conduct standard content analysis and systematic comparison of data between the two intervention groups; acceptability, appropriateness, patterns in facilitators/barriers, implementation quality, and early sustainment.

In sum, these interviews will provide more in-depth understanding of the ethical implications of our intervention and evaluation of the implementation process by relevant stakeholders.

ELIGIBILITY:
Proband Inclusion Criteria:

* KCNQ1 Thr224Met or APOB R3527Q carrier
* 18 years or older

Proband Exclusion Criteria:

* None

Family Inclusion Criteria:

* 1st degree relative of a KCNQ1 Thr224Met or APOB Arg3527Gln carrier

Family Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Uptake of cascade screening among all first-degree relatives | Through study completion: approximately 4 years
  Proportion of first-degree relatives who undergo testing/All eligible first-degree relatives

SECONDARY OUTCOMES:
Number of new cases detected among all first-degree family members | Through study completion: approximately 4 years
  New cases/All eligible first-degree family members
Perceived alignment of ethical principles questionnaire | up to 6 months
  Among probands and family members
Anxiety regarding method of contact questionnaire | up to 6 months
  Among probands and family members
Perceived pressure to undergo testing/share health information questionnaire | up to 6 months
  Among probands and family members
Knowledge of disease and variant questionnaire | up to 6 months
  Among probands and family members

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No